CLINICAL TRIAL: NCT00233597
Title: A Phase III Study of the Safety and Efficacy of Ferumoxytol (Compared With Oral Iron) as an Iron Replacement Therapy in Hemodialysis Patients Who Are Receiving Supplemental EPO Therapy
Brief Title: Ferumoxytol Versus Oral Iron in the Treatment of Anemia in Hemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 62745-5
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Anemia
Keywords: anemia; iron
MeSH Terms: conditions — Anemia | interventions — Ferrosoferric Oxide; Iron

INTERVENTIONS:
Drug: ferumoxytol or oral iron

SUMMARY:
The study will evaluate the safety and efficacy of a new intravenously administered iron drug to treat anemia in patients on hemodialysis.

DETAILED DESCRIPTION:
This study will evaluate the efficacy and safety of intravenous (IV) iron (ferumoxytol) as compared to oral iron in the treatment of anemia in hemodialysis patients receiving erythropoietin. Patients are randomized to receive either two doses of 510 mg of intravenous ferumoxytol in sequential dialysis sessions or 200 mg oral elemental iron daily for three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years.
* Chronic hemodialysis.
* Stable supplemental EPO therapy.
* Baseline hemoglobin of ≤ 11.5 g/dl.

Exclusion Criteria:

* Women who are pregnant or who are breast feeding.
* Received another investigational drug or device within 30 days.
* Recent parenteral or oral iron therapy.
* Patients with active GI bleeding or acute bleeding within 4 weeks. Patients that have other causes of anemia.
* Major surgery within 30 days or anticipated or planned surgery during the study.
* Patients with active infections.
* Recent blood transfusions.
* Patients with known allergies to iron products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230
Dates: Start 2004-08; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The mean change in hemoglobin from baseline.

SECONDARY OUTCOMES:
Change in iron indices.

CONTACTS AND LOCATIONS:
Locations (45):
- United States (45):
  - Phoenix, Arizona
  - Tempe, Arizona
  - Los Angeles, California
  - Mountain View, California
  - New Haven, Connecticut
  - Hudson, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Honolulu, Hawaii
  - Gurnee, Illinois
  - Hines, Illinois
  - Baton Rouge, Louisiana
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Columbus, Mississippi
  - Jackson, Mississippi
  - Kansas City, Missouri
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Flushing, New York
  - Mineola, New York
  - New York, New York
  - Orchard Park, New York
  - Springfield Gardens, New York
  - Chapel Hill, North Carolina
  - Portland, Oregon
  - Lewistown, Pennsylvania
  - Greenville, South Carolina
  - Sumter, South Carolina
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - Alexandria, Virginia
  - Chesapeake, Virginia
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Salem, Virginia
  - Spokane, Washington
  - Appleton, Wisconsin

REFERENCES:
- [Background] Landry R, Jacobs PM, Davis R, Shenouda M, Bolton WK. Pharmacokinetic study of ferumoxytol: a new iron replacement therapy in normal subjects and hemodialysis patients. Am J Nephrol. 2005 Jul-Aug;25(4):400-10. doi: 10.1159/000087212. Epub 2005 Jul 28. PMID 16088081
- [Result] Provenzano R, Schiller B, Rao M, Coyne D, Brenner L, Pereira BJ. Ferumoxytol as an intravenous iron replacement therapy in hemodialysis patients. Clin J Am Soc Nephrol. 2009 Feb;4(2):386-93. doi: 10.2215/CJN.02840608. Epub 2009 Jan 28. PMID 19176796
- See also: National Kidney Foundation — http://www.kidney.org/index.cfm